CLINICAL TRIAL: NCT00637455
Title: Single Center, Randomized,Double-Blind,Crossover Study Comparing the Effects of Single-Dose Fexofenadine HCl 180 mg, Cetirizine 10 mg, and Placebo on Cognitive Performance in Naval Flight Personnel
Brief Title: Single Center, Randomized, Double-Blind,Crossover Study Comparing Effects Of Single-Dose Fexofenadine HCl 180 mg, Cetirizine 10 mg, and Placebo on Cognitive Performance in Naval Flight Personnel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A/4139
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — fexofenadine

INTERVENTIONS:
Drug: fexofenadine HCl
  Other Names: Allegra

SUMMARY:
To compare the effects of fexofenadine HCl 180 mg, cetirizine 10 mg, and placebo on computerized scores derived from the Aeromedical Vigilance Task (AVT), a computerized objective measure of attention, accuracy and reaction time in healthy naval flight personnel. Specifically, the primary objective is to compare the AVT overall (average of the 18 blocks) mean change from baseline in total number of errors (commission errors + omission errors) between fexofenadine HCl and cetirizine 10 mg. Safety of these single-dose treatments also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female naval flight personnel, ≥18 years of age
* CogScreen-AE Logistic Regression Probability Value < 0.6 at the baseline screening visit
* Normal SaO2 (>95%) as measured by pulse oximetry
* Female subjects must be of nonchildbearing potential (i.e., surgically sterile or at least 1 year postmenopausal); see Section 4.4 for additional information:

Exclusion Criteria:

* Female subjects who are pregnant, lactating, or likely to become pregnant during the study
* Signs or symptoms of currently active allergic disease (seasonal allergic rhinitis, perennial allergic rhinitis, episodic allergic rhinitis) within 2 weeks prior to the screening visit
* Upper respiratory tract infection, sinusitis, asthma exacerbation, or flu-like symptoms within 2 weeks prior to the screening visit
* Medical history or physical examination findings; clinically significant cardiovascular, respiratory, hepatic, neurologic, endocrine, psychiatric, or other major systemic disease; or laboratory or electrocardiograph abnormality making implementation of the protocol or interpretation of the protocol results difficult. Abnormalities which are not clinically significant will not necessarily disqualify subjects provided, in the opinion of the investigator and sponsor, the study validity or the subject's welfare is not compromised.
* Any unusual sleep pattern, including third-shift workers (11:00 PM to 7:00 AM), or sleep < 6 hours the night before each AVT testing at Visits 1-4
* Any excessive amounts of alcohol (no more than two drinks/day on average)
* Any excessive use of caffeine (more than three cups of coffee per day or equivalent)
* Any history of chronic alcohol or mood-altering drug abuse
* Any use of tobacco/nicotine products within 90 days of the screening visit or during the study
* Any disease state or surgery known to affect the gastrointestinal absorption of drugs
* Mental capacity limited to the extent the subject cannot give legal informed consent or accurate information regarding efficacy and side effects/tolerance of drug
* Subjects unable to comply with the protocol requirements (must complete a screening visit and Visits 1-4 within approximately 1-1/2 months)
* Known hypersensitivity to fexofenadine, or the tablet ingredients (croscarmellose sodium, magnesium stearate, microcrystalline cellulose, pregelatinized starch; or the tablet coating made of hydroxypropyl methylcellulose, iron oxide blends, polyethylene glycol, povidone, silicone dioxide, and titanium dioxide)
* Known hypersensitivity to cetirizine or the tablet ingredients (lactose, magnesium stearate, povidone, titanium dioxide, hydroxypropyl methylcellulose, polyethylene glycol, and corn starch)
* Use of an investigational drug within 30 days prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-09; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Compare the AVT overall mean challenge from baseline between Fexofenadine HCl & Cetirizine

SECONDARY OUTCOMES:
Evaluating change from baseline between Fexofenadine HCl and Cetirizine on the endpoint of total # of errors under each normobaric hypoxic condition

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States